CLINICAL TRIAL: NCT02787122
Title: Comparison of Emotion-focused Cognitive Behavior Therapy for Patients With Schizophrenia With Standard Treatment: Effects on Psychological Parameters and Rehospitalisation
Brief Title: Pilot-trial of Emotion-focused Cognitive Behavior Therapy for Patients With Schizophrenia
Acronym: CBT-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stephanie Mehl, Prof. Dr. rer. nat., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT-E_MehlLincoln
Record Dates: First submitted 2016-03-03; First posted 2016-06-01 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia; Delusional Disorder; Schizoaffective Disorder; Brief Psychotic Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; psychotic disorders; Cognitive Behavior Therapy; emotion regulation; self-esteem; randomized-controlled trial
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Paranoid; Psychotic Disorders; Emotional Regulation | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The CBT-E group receives 15-25 sessions of cognitive behavior therapy with a special focus on emotion regulation (CBT-E), the wait list group receives CBT-E after six month waiting time
Who Masked: Participant
Masking Description: Blinded rating of diagnostic interviews
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-E (Active Comparator): Emotion-focussed Cognitive behavior therapy:
  Patients receive 25 sessions of individual emotion-focused Cognitive Behavior Therapy. Interventions are behavioral activation, training of emotion regulation strategies, improvement of self-esteem and relapse prevention.
  Interventions: Behavioral: CBT-E
- Treatment as Usual (Placebo Comparator): Patients who are randomized and assigned to the Wait list are required to wait for half a year, while they receive standardized care (antipsychotic medication). After half a year, they receive CBT-E, as well.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: CBT-E — Patients receive 25 sessions of individual emotion-focused Cognitive Behavior Therapy based on a manual. Interventions aim on patients' mood by implementing positive activities in their daily routine. Further, patients train to reduce worrying behavior. Social contacts are fostered as well. Later, patients are informed on emotions and train emotion regulation strategies. Finally, the focus of CBT-E is on self-acceptance.Patients receive psychoeducation on self-acceptance and learn strategies in order to reduce negative self-schema and foster positive self-schema.
  Other Names: Emotion-focused Cognitive Behavior Therapy
  Arms: CBT-E
Behavioral: Treatment as Usual — Patients receive standardized treatment. After a waiting period of six month, patients receive CBT-E
  Arms: Treatment as Usual

SUMMARY:
The present study is a pilot single-blind randomized controlled therapy study. Its aim is to assess the efficacy of an emotion-focussed form of Cognitive behavior Therapy that focusses on emotional processes that are involved in the formation and maintenance of delusions such as emotional stability, emotion regulation and self-esteem.

DETAILED DESCRIPTION:
Cognitive Behavior Therapy for psychosis (CBTp) is an effective treatment for patients with psychosis. Several meta-analyses showed an effect of CBTp in addition to antipsychotic treatment of small to medium effect size with regard to positive symptoms, general psychopathology and depression. Nevertheless, present research suggests that are especially emotional processes are closely related to positive symptoms and delusions, such as negative emotions, low self-esteem, depression and anxiety, whereas present interventions of CBTp focus often especially on cognitive interventions in order to change delusions as well as more cognitive risk factors for delusions such as reasoning biases and a dysfunctional causal attribution style.

Thus, the aim of the present single-blind randomized-controlled pilot therapy study was to assess the efficacy of a new form of emotion-focussed Cognitive behavior therapy for psychosis with regard to change in positive symptoms and delusions in comparison to standard treatment.

The main hypotheses are:

- Efficacy of CBT-E: patients with schizophrenia who receive CBT-E show a more pronounced reduction of delusions (primary outcome), as well as a more pronounced reduction of positive symptoms, depression and general psychopathology, a stronger improvement in general and social functioning and will receive lower doses of antipsychotic medication (secondary outcomes) at post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, delusional disorder or brief psychotic disorder
* Positive and Negative Syndrome Scale score in item P1 (delusions) of at least two
* fluent in German language
* agree to participate
* estimated general intelligence of at least 70 (assessed with the German Wortschatztest (MWT-B)
* no present suicidality

Exclusion Criteria:

* acute suicidality
* comorbid diagnosis of borderline personality disorder and/or substance use disorder in the last six month
* intake of Benzodiazepines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Psychotic Rating Scale (PSYRATS) delusions scale | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of delusion frequency, delusion distress, conviction and loss of quality of life

SECONDARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of positive, negative and general symptoms of schizophrenia
Change in Calgary Depression Rating Scale for Schizophrenia (CDSS) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of depressive symptoms in patients with schizophrenia
Change in Role Functioning Scale (RFS) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of social functioning
Change in Paranoia Checklist (PCL) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of self-reported paranoid delusion frequency, distress and conviction
Change in Beck Depression Inventory-II | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of self-reported depressive symptoms
Change in Peters et al. Delusions Inventory | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of self-rated delusion frequency, delusional distress and delusional

OTHER OUTCOMES:
Change in Reactions to paranoid thoughts Scale (REPT) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of cognitive and emotional reactions on paranoid thoughts
Change in Symptom Checklist 9 (SCL-9) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of severity of self-reported symptoms of different mental disorders (depression, anxiety, phobia, obsessive-compulsive symptoms, etc.)
Change in Satisfaction With Life Scale (SWLS) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of life satisfaction
Change in Pittsburg Sleep Quality Inventory (PSQI) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of objective sleep quality and sleep problems
Change in number of social contacts (SozE) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of number of social contacts in the last week
Change in Perseverative Thinking Questionnaire (PTQ) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of self-reported perseverative thinking and worrying
Change in Scale of Emotion Regulation Competencies (SEK-27) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of self-reported habitual use of different emotion regulation strategies
Change in Self-Compassion Scale (SCS) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of self-reported self-compassion
Change in Brief Core Schema Scale (BCSS) | Change between assessment pre-therapy and assessment after six month of therapy
  Assessment of positive and negative self-schemas and positive and negative schemas of other persons

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Mehl, Ph. D., Principal Investigator — Philipps University Marburg; Tania M. Lincoln, Principal Investigator — University of Hamburg-Eppendorf; Winfried Rief, Study Director — Philipps University Marburg; Tilo Kircher, Study Director — Philipps University Marburg
Locations (2):
- Germany (2):
  - University of Marburg, Faculty of Clinical Psychology and Psychotherapy, Marburg, Hesse
  - University of Hamburg, Faculty of Clinical Psychology and Psychotherapy, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided